CLINICAL TRIAL: NCT02246842
Title: A Randomised Study Comparing the Pharmacokinetics and Tolerance of D-Gam® 1500IU to Rhophylac® 1500IUin Rh-D-negative Healthy Volunteers.
Brief Title: A Study Comparing the Pharmacokinetics and Tolerance of D-Gam® to Rhophylac® in Rh-D-negative Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bio Products Laboratory (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: POLYAD04
Record Dates: First submitted 2014-09-15; First posted 2014-09-23 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Healthy
Keywords: Volunteers
MeSH Terms: interventions — Rho(D) Immune Globulin

ARMS (2):
- D-Gam® (Experimental): D-Gam® (human anti-D immunoglobulin)
  Interventions: Biological: D-Gam® (human anti-D immunoglobulin)
- Rhophylac® (Active Comparator): Human Anti-D Immunoglobulin
  Interventions: Biological: Rhophylac® (human anti-D immunoglobulin)

INTERVENTIONS:
Biological: D-Gam® (human anti-D immunoglobulin)
  Arms: D-Gam®
Biological: Rhophylac® (human anti-D immunoglobulin)
  Arms: Rhophylac®

SUMMARY:
The primary objective of the study was to compare peak serum anti-D levels (Cmax) of BPL's D-Gam® 1500 IU to Rhophylac® 1500IU in RhD-negative healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Females
* Ages of 18 and 55 years
* Bodyweight of 50-85kg.

Exclusion Criteria:

* Clinically relevant abnormalities at physical examination, ECG or laboratory tests.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-05; Primary Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Cmax for anti-D | Pre-dose, 1, 8, 24, 32, 48, 72 & 96 hours; 1, 2, 3, 4, 5, 6, 8, 10, 12 & 14 weeks post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Dr A Sutton, MB BS, FFARCSI, Principal Investigator — Guildford Clinical Pharmacology Unit
Locations (1):
- Guildford Clinical Pharmacology Unit, Unit 34, Surrey Technology Centre, Surrey Research Park, Occam Road, Guildford, Surrey, United Kingdom

REFERENCES:
- See also: Sponsor's Homepage — http://www.bpl.co.uk